CLINICAL TRIAL: NCT07121153
Title: Investigation of Safety, Tolerability and Pharmacokinetic Properties of Single Doses of Subcutaneous NNC0487-0111 in Chinese Participants With Overweight or Obesity.
Brief Title: A Research Study on How NNC0487-0111, a New Medicine, Works in Chinese Participants When Injected Under the Skin.
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: NN9490-8213; U1111-1311-5582 (Other: WHO)
Record Dates: First submitted 2025-08-07; First posted 2025-08-13 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort A1 (Experimental): Cohort A1 will include 12 participants randomised (3:1), with 9 participants being randomised to receive a single dose level 1 of active treatment and 3 participants randomised to receive placebo.
  Interventions: Drug: NNC0487-0111 A; Drug: Placebo A
- Cohort A2 (Experimental): Cohort A2 will include 12 participants randomised (3:1), with 9 participants being randomised to receive a single dose level 2 of active treatment and 3 participants randomised to receive placebo.
  Interventions: Drug: NNC0487-0111 A; Drug: Placebo A
- Cohort A3 (Experimental): Cohort A3 will include 12 participants randomised (3:1), with 9 participants being randomised to receive a single dose level 3 of active treatment and 3 participants randomised to receive placebo.
  Interventions: Drug: NNC0487-0111 A; Drug: Placebo A

INTERVENTIONS:
Drug: NNC0487-0111 A — Participants will receive single dose (level 1, level 2, level 3) injection of NNC0487-0111 A subcutaneoulsy.
Drug: Placebo A — Participants will receive single dose (level 1, level 2, level 3) injection of placebo A subcutaneoulsy.

SUMMARY:
The study is testing a new medicine (NNC0487-0111) for weight control in Chinese people with BMI between 24 kilogram per meter square (kg/m2) and 34.9 kg/m2. The aim of the study is to see how safe the study medicine is and how it behaves in human body. Participants will either get the study medicine or placebo (a "dummy medicine" similar to the study medicine but without active ingredients) and which treatment they get is decided by chance. The study medicine is a potential new medicine which cannot be prescribed by doctors but has previously been tested in humans. This study will last for up to 53 days.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent obtained before any study-related activities. Study-related activities are any procedures that are carried out as part of the study, including activities to determine suitability for the study.
2. Male Chinese participants, age 18-55 years (both inclusive) at the time of signing the informed consent.
3. Body mass index between 24.0 and 34.9 kg/m2 (both inclusive) at screening. Overweight and obesity should be due to excess adipose tissue, as judged by the investigator, with a body weight (more than or equal to) ≥ 65.0 kg at screening.
4. Considered eligible based on the medical history, physical examination, and the results of vital signs, electrocardiogram and clinical laboratory tests performed during the screening visit, as judged by the investigator.

Exclusion Criteria:

1. Any condition, unwillingness or inability which in the investigator's opinion might jeopardise participant's safety or compliance with the protocol.
2. HbA1c ≥ 6.5 percent (%) [48 milimol per mole (mmol/mol)] at screening.
3. Any laboratory safety parameters at screening outside the below laboratory ranges:

   * Vitamin D (25-hydroxycholecalciferol) less than (<) 12 nanogram per mililiter (ng/mL) [30 nanometer (nM)] at screening
   * Parathyroid hormone (PTH) outside normal range at screening
   * Total calcium outside normal range at screening
   * Amylase ≥ 2 times upper limit of normal at screening
   * Lipase ≥ 2 times upper limit of normal at screening
   * Calcitonin ≥ 50 picogram per mililiter (pg/mL) at screening

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-08-11 (Actual); Primary Completion 2026-01-11 (Estimated); Study Completion 2026-01-11 (Estimated)

PRIMARY OUTCOMES:
Number of treatment emergent adverse events (TEAEs) | From NNC0487-0111 administration (Day 1) to completion of the end of study visit (Day 23)
  Number of events

SECONDARY OUTCOMES:
AUC0-∞,SD; the area under the NNC0487-0111 plasma concentration-time curve from time 0 to infinity after a single dose | From pre-dose on Day 1 until completion of the end of study visit (Day 23)
  h*nmol/L
Cmax,SD; the maximum plasma concentration of NNC0487-0111 after a single dose | From pre-dose on Day 1 until completion of the end of study visit (Day 23)
  nmol/L
tmax,SD; the time of maximum plasma concentration of NNC0487-0111 after a single dose | From pre-dose on Day 1 until completion of the end of study visit (Day 23)
  h
t1/2,SD; the terminal half-life of NNC0487-0111 after a single dose | From pre-dose on Day 1 until completion of the end of study visit (Day 23)
  h
Relative change in body weight | From baseline Day 1 until completion of the end of study visit (Day 23)
Change in fasting plasma glucose | From baseline Day 1 until completion of the end of study visit (Day 23)
  mmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency dept. 2834, Study Director — Novo Nordisk A/S
Locations (1):
- Jinan Central Hospital Affiliated to Shandong University, Ji'Nan, Shandong, China

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://novonordisk-trials.com